CLINICAL TRIAL: NCT06573853
Title: The Safety and Efficiency of Pulsed Field Ablation and Radiofrequency Ablation in the Treatment of Paroxysmal Supraventricular Tachycardia：a Retrospective and Propensity Score Matching Study
Brief Title: Outcomes of PFA Vs. RFA for Patients with PSVT: a Retrospective and Propensity Score Matching Study
Acronym: PFA*RFA*PSVT
Status: Recruiting | Type: Observational
Sponsor: Caijie Shen (Other)
Collaborators: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Caijie Shen, Associate Chief Physician of the First Affiliated Hospital of Ningbo University, Ningbo No. 1 Hospital
Organization: Ningbo No. 1 Hospital (Other)
Other Study IDs: 775050
Record Dates: First submitted 2024-08-09; First posted 2024-08-27 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Supraventricular Tachycardia; Catheter Ablation
Keywords: Paroxysmal Supraventricular Tachycardia; Pulsed Field Ablation; Radiofrequency Ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PFA group: A retrospective analysis was conducted on 214 patients with PSVT recieving PFA who met the inclusion and exclusion criteria and visited at the First Affiliated Hospital of Ningbo University, the Third People's Hospital of Chengdu, the Xiamen Cardiovascular Hospital of Xiamen University, the First Hospital of Jilin University, the Seventh People's Hospital of Zhengzhou, Shanghai General Hospital, and Jiangxi Provincial People's Hospital from October 2022 to June 2024. These patients were included in the PFA group. Basic clinical information, procedural data, and the efficiency and safety post 1-year follow-up were collected and analyzed.
  Interventions: Procedure: Focal Pulsed Field Ablation (PFA)
- RFA group: A retrospective analysis for control group was conducted on patients with PSVT reciecing RFA who met the inclusion and exclusion criteria and visited at the First Affiliated Hospital of Ningbo University the Third People's Hospital of Chengdu, the Xiamen Cardiovascular Hospital of Xiamen University, the First Hospital of Jilin University, the Seventh People's Hospital of Zhengzhou, Shanghai General Hospital, and Jiangxi Provincial People's Hospital from October 2022 to June 2024. 214 patients approached by RFA were matched 1:1 by propensity score to a similar population treated by PFA. Basic clinical information, procedural data, as well as the efficiency and safety of 1-year follow-up were collected and analyzed.
  Interventions: Procedure: Focal Radiofrequecy Ablation (RFA)

INTERVENTIONS:
Procedure: Focal Pulsed Field Ablation (PFA) — Patients in the PFA group underwent ablation procedures utilizing a force-sensing PFA catheter for the treatment of PSVT.
  Groups: PFA group
Procedure: Focal Radiofrequecy Ablation (RFA) — Patients in the PFA group underwent ablation procedures utilizing force-sensing RFA catheters for the treatment of PSVT.
  Groups: RFA group

SUMMARY:
The goal of this retrospective study is to compare the long-term follow-up outcomes of pulses field ablation (PFA) Vs. radiofrequency ablation (RFA) for the patients with paroxysmal supraventricular tachycardia (PSVT). The main question to answer is:

Does the PFA was more effecient and safer that RFA for treatment of PSVT during procedure and after 1-year follow-up? Researchers will compare the acute and long-term efficiency and safety between PFA and RFA.

1. Recieved PFA or RFA 1 year ago
2. Finish the visit to the clinic at 1, 3, 6, 12 months for examinations and blood testings
3. Patients recieved PFA and PFA under propensity matched comparison according to differen variety of PSVT

DETAILED DESCRIPTION:
The goal of this retrospective study is to compare the long-term follow-up outcomes of PFA Vs. RFA for the patients with PSVT. The main question to answer is:

Does the PFA was more effecient and safer that RFA for treatment of PSVT during procedure and after 1-year follow-up? Researchers will compare the acute and long-term efficiency and safety between PFA and RFA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic PSVT including: atrioventricular nodal re-entrant tachycardia (AVNRT), atrioventricular re-entrant tachycardia (AVRT);
2. Age range: 18 years old ≤ age ≤ 80 years old, with no gender restriction;
3. Willing to receive the examinations and testings during one year follow-up required by the protocol;
4. Voluntary signed informed consent.

Exclusion Criteria:

1. Organic heart disease;
2. History of cardiac surgery;
3. Previous failed ablation of PSVT;
4. Presence of any implants, such as a permanent pacemaker;
5. Patients with invasive systemic infections or advanced malignant tumors;
6. Contraindications for septal puncture or retrograde transaortic access surgery;
7. Any condition that makes the use of heparin or aspirin inappropriate;
8. Pregnant or lactating women;
9. Inability to fully comply with the study procedures and follow-ups or to provide their own informed consent;
10. Coexistence with other arrhythmias, such as atrial fibrillation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PSVT was documented with a 12-lead surface electrocardiogram (ECG), 24-hour Holter monitoring, and esophageal electrophysiologic study (EES) before hospitalization. A diagnosis of AVNRT or AVRT was confirmed by electrophysiological study after the antiarrhythmic medications were withdrawn ≥5 half-lives. Patients with reproducibly clinical PSVT were finally enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute and long-term follow-up success rate | 15 minutes post ablation for acute sussess and one year for follow-up success
  The Primary endpoints for efficacy included the number of subjects with acute and long-term follow-up success post ablation. The acute success was confirmed by noninducibility of clinical PSVT after programmed stimuli and drug administration after15 minutes waiting time. The long-term follow-up success was defined as the absence of clinical PSVT during the 1-year follow-up.
  The acute success is confirmed by catheter mapping and ECG to determine immediate ablation success rate
Incidence of intraoperative and long-term serious adverse events | 24 hours post ablation for intraoperative serious adverse events and one year for follow-up serious adverse events
  The Primary endpoints for safety included the number of subjects suffering from serious adverse events. The incidence of serious adverse events related to the ablation included conduction system impairment, ventricular arrhythmia, myocardial infarction, hemolysis or major bleeding requiring transfusion, cardiac tamponade/perforation, Pericarditis requiring treatment, infectious endocarditis, valve stenosis or regurgitation deterioration, heart failure, abnormal renal and/or hepatic function, Intracerebral hemorrhage/transient ischemic attack/ stroke, and death. (Abnormal renal function (dialysis, transplant, serum creatinine >200 mmol/L); Abnormal hepatic function (cirrhosis, bilirubin > x 2 upper limit of normal, aspartate aminotransferase/alkaline phosphatase/alanine aminotransferase >3 x upper limit of normal).

SECONDARY OUTCOMES:
Non-serious adverse events | 24 hours post ablation for intraoperative serious adverse events and 1 year for follow-up serious adverse events
  Muscle constraction delaying the procedure, untolerable pain or cough, abnormal renal function (without dialysisserum, creatinine <200 mmol/L), and abnormal hepatic function (cirrhosis, bilirubin < x 2 upper limit of normal, aspartate aminotransferase/alkaline phosphatase/alanine aminotransferase <3 x upper limit of normal.

CONTACTS AND LOCATIONS:
Overall Officials: Caijie Shen, Study Director — First Affiliated Hospital of Ningbo University
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen C, Jia Z, Yu Y, Feng M, Du X, Fu G, Yu L, Wu T, Jiang Y, Jin H, Zhuo W, Gao F, Wang B, Chen S, Dai J, Fang R, Chu H. Efficacy and safety of pulsed field ablation for accessory pathways: a pilot study. Europace. 2024 Jul 2;26(7):euae139. doi: 10.1093/europace/euae139. PMID 38801673
- [Background] Shen C, Du X, Dai J, Feng M, Yu Y, Liu J, Fu G, Wang B, Jiang Y, Jin H, Chu H. Outcomes of Focal Pulsed Field Ablation for Paroxysmal Supraventricular Tachycardia. Can J Cardiol. 2024 Jul;40(7):1294-1303. doi: 10.1016/j.cjca.2023.12.037. Epub 2024 Jan 17. PMID 38242530